CLINICAL TRIAL: NCT03979222
Title: Observational Cohort Study of a National Extracorporeal Membrane Oxygenation Service for Adults With Respiratory Failure: the NHS ECMO Study.
Acronym: NHS ECMO
Status: Completed | Type: Observational
Sponsor: University of Cambridge (Other)
Collaborators: Royal Papworth Hospital Clinical Trials Unit (Unknown); Aberdeen Royal Infirmary, NHS Grampian (Unknown); Guy's and St Thomas' NHS Foundation Trust (Other); Royal Brompton & Harefield Hospitals NHS Foundation Trust (Unknown); Royal Papworth Hospital NHS Foundation Trust (Unknown); University Hospitals of Leicester NHS Foundation Trust (Unknown); Manchester University NHS Foundation Trust (Other Government); NHS England (Other Government)
Responsible Party: Principal Investigator, Alex Warren, Academic Foundation Doctor, Division of Anaesthesia, University of Cambridge
Other Study IDs: ECMO-001
Record Dates: First submitted 2019-06-02; First posted 2019-06-07 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Acute Respiratory Failure
Keywords: ECMO; ARDS; Acute respiratory failure
MeSH Terms: interventions — Extracorporeal Membrane Oxygenation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Extracorporeal Membrane Oxygenation — ECMO provides extracorporeal gas exchange through use of a membrane oxygenator. Blood is drained from a central vein and returned after oxygenation into either the venous or arterial circulation dependent on configuration.

SUMMARY:
This is an observational study of outcomes of the NHS England-commissioned national respiratory ECMO service, which has been active at six centres since December 2011.

The primary outcome of interest is the number of patients who survive to ICU discharge at the ECMO centre. The study also aims to identify factors predictive of outcome.

DETAILED DESCRIPTION:
Recent randomised and observational studies suggest there may be a role for extracorporeal membrane oxygenation (ECMO) in patients with severe acute respiratory failure that have not responded to conventional measures.

In 2011, NHS England commissioned a national service to provide ECMO for severe respiratory failure at six centres across the country. Patients with severe respiratory failure are referred to the network if conventional measures are unsuccessful, and if accepted are transferred to an ECMO centre for specialist care. The criteria for admission is at the discretion of clinicians at each centre.

The NHS ECMO registry has been created by cross-referencing data submitted to the Extracorporeal Life Support Organisation (ELSO) in Ann Arbor, Michigan, with a tracker document identifying patients treated within the network. Analysis has been undertaken from December 2018 to March 2019.

ELIGIBILITY:
Inclusion Criteria:

* Ultimately at the discretion of the clinician at the relevant ECMO centre
* Aged ≥16 years
* Severe acute respiratory failure refractory to conventional management
* No contra-indication to ongoing ECMO therapy

Exclusion Criteria:

* Any contra-indication to ongoing ECMO therapy
* Need for ECMO due to other aetiology than acute respiratory failure (e.g. bridge to transplantation, extracorporeal CPR, isolated acute cardiac failure)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who received ECMO as part of the NHS England-commissioned national respiratory ECMO service between 1st December 2011 and 31st December 2017.
Sampling Method: Non-Probability Sample
Enrollment: 1205 (Actual)
Dates: Start 2011-12-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Survival at ECMO ICU discharge | Up to 90 days.
  The proportion of patients who are alive at discharge from the ICU at the treating ECMO centre.

SECONDARY OUTCOMES:
Duration of ECMO treatment. | Up to 90 days.
  The time (hours) where the patient is actively supported by the ECMO circuit.
Frequency of Complications | Up to 90 days.
  The proportion of patients experiencing recognised complications of ECMO treatment.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Warren A, Chiu YD, Villar SS, Fowles JA, Symes N, Barker J, Camporota L, Harvey C, Ledot S, Scott I, Vuylsteke A; NHS England-commissioned National ECMO Service. Outcomes of the NHS England National Extracorporeal Membrane Oxygenation Service for adults with respiratory failure: a multicentre observational cohort study. Br J Anaesth. 2020 Sep;125(3):259-266. doi: 10.1016/j.bja.2020.05.065. Epub 2020 Jul 28. PMID 32736826

DOCUMENTS (1):
  • Statistical Analysis Plan (2019-02-25): https://cdn.clinicaltrials.gov/large-docs/22/NCT03979222/SAP_000.pdf